CLINICAL TRIAL: NCT03540680
Title: Case-control Study Evaluating the Impact of p16Ink4a in Bronchopulmonary Dysplasia in Children
Brief Title: p16Ink4a in Bronchopulmonary Dysplasia in Children
Acronym: DBP16
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DBP16
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Term newborns (≥37GA) (Other): Blood punction on the cordon
  Interventions: Other: Blood punction
- Premature newborns (Other): Blood punction on the cordon
  Interventions: Other: Blood punction
- Child between 7 and 15 years old with BPD (Other): Blood punction
  Interventions: Other: Blood punction
- Child between 7 and 15 years old without BPD (Other): Blood punction
  Interventions: Other: Blood punction

INTERVENTIONS:
Other: Blood punction — For the arms "Term newborns (≥37GA)" and "Premature newborns" the only intervention is a blood punction on the cordon.
  For the arms "Child between 7 and 15 years old" with or without BPD the only intervention is a blood punction on peripheral blood.

SUMMARY:
The bronchopulmonary dysplasia (BPD) is a respiratory disease of the premature child which lead to a reduction of gas exchange surface and to a prolonged respiratory failure. This disease has morphologic and functional consequences at adulthood and is today considered to be an early determinant of respiratory diseases at adulthood.

The physiopathology of BPD is not well known. Several mechanisms could be involved especially a reparation failure favored by an increase of cellular senescence which is a permanent stop of cellular proliferation. The transcription factor 16 Ink4a, considered as a marker of aging, is one of the essential markers of senescence. Its increase during prematurity was shown at the blood cells of the cordon, but its involvement in BPD and its evolution in child are not yet studied.

ELIGIBILITY:
Inclusion Criteria:

Premature(< 28 GA) neonates

* Alive neonate born at less than 28 gestational age
* Signed inform consent

Term neonates:

* Alive neonate born at least at 37 GA or more
* Signed inform consent

Child from 7 to 15 years old with BPD:

* Child from 7 to 15 years old
* Child with a BPD diagnosed
* Signed inform consent

Child from 7 to 15 years old without BPD:

* Child from 7 to 15 years old
* Child receiving a blood test
* Signed inform consent

Exclusion Criteria:

Premature (< 28 GA) and term neonates:

-Congenital malformation

Child from 7 to 15 years old with BPD:

* Cystic fibrosis
* Evolutive cancer
* Chronic inflammatory disease
* Known anemia
* Refusal of participation of child or parental authority

Child from 7 to 15 years old without BPD:

* Other respiratory disease: severe asthma, cystic fibrosis, deficit AAT, bronchial dilatation
* Evolutive cancer
* Chronic inflammatory disease
* Known anemia
* Refusal of participation of child or parental authority

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
p16 expression | Day 1
  p16 expression measured by qPCR in newborns cord blood cells and in circulating leukocytes of children aged from 7 to 15

SECONDARY OUTCOMES:
Telomeres length | Day 1
  Telomeres length of circulating leukocytes
Genetic expression of p21, p53, H2Ax | Day 1
  Genetic expression of p21, p53, H2Ax of circulating leukocytes

CONTACTS AND LOCATIONS:
Overall Officials: Ralph EPAUD, MD, Principal Investigator — CHI Créteil
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France